CLINICAL TRIAL: NCT00704210
Title: Effectiveness of Mechanical Decompression for Low Back Pain Relief
Acronym: SpiDERS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn by sponsor
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, William Grant, Professor, Family Medicine, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRBPHS 5379
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Sham Comparator): Group B will receive sham decompression treatment (i.e. tension not exceeding 15 lbs) for 30 minutes and ice treatment for 15 minutes once a day during each treatment session. No incremental increases will be used for Group B.
  Interventions: Device: SpineMed Table, Cert HealthSciences LLC
- A (Experimental): For Group A (the treated group) the following tension adjustments will be used: starting treatment tension will equal 1/4 body weight minus 10 lbs. Incremental increases of 4 lbs. per session will be implemented until optimum tensions are reached, which would be a maximum of ¼ body weight plus 25 lbs, unless distraction tensions cause discomfort, which would require a reduction of the tensions applied.
  Interventions: Device: SpineMed Table, Cert HealthSciences LLC

INTERVENTIONS:
Device: SpineMed Table, Cert HealthSciences LLC — For Group A (the treated group) the following tension adjustments will be used: starting treatment tension will equal 1/4 body weight minus 10 lbs. Incremental increases of 4 lbs. per session will be implemented until optimum tensions are reached, which would be a maximum of ¼ body weight plus 25 lbs, unless distraction tensions cause discomfort, which would require a reduction of the tensions applied.
  Arms: A
Device: SpineMed Table, Cert HealthSciences LLC — Group B will receive sham decompression treatment (i.e. tension not exceeding 15 lbs) for 30 minutes and ice treatment for 15 minutes once a day during each treatment session. No incremental increases will be used for Group B.
  Arms: B

SUMMARY:
Objective To demonstrate the effectiveness of a conservative treatment approach for chronic low back pain that addresses the underlying problem of intervertebral disc lesions and degenerative disc disease, namely vertebral pressure on vital structures of the lumbar region.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common medical problem and a challenging condition to treat. This study will investigate the effectiveness of a conservative treatment approach for chronic LBP. To this point few treatment approaches specifically address the resolution of underlying pathologies leading to a high probability of recurrence of LBP. Further, current treatment options for lumbar disc pathology have been of limited demonstrated effectiveness. The purpose of this study is to determine whether a non-surgical therapeutic approach designed to effect intervertebral widening and allow for reduction of disc protrusion will reduce patients' pain and improve their activity levels.

The study will assess whether a computer-assisted traction treatment [decompression] protocol results in improvement in patient pain levels and daily activity levels. Further, to determine if such treatment results in intervertebral widening and reduction of any disc protrusions as demonstrated by direct imaging of the lumbar spine. A double-blind (treatment vs. sham treatment) design will be employed

Specific Aims To study the effectiveness of decompression therapy for LBP patients with lumbar disc herniation and degenerative disc problems.

To demonstrate that decompression therapy for LBP patients results in a demonstrated reduction in levels of reported pain.

To demonstrate that decompression therapy for LBP patients results in a demonstrated greater return to daily activities.

To demonstrate that decompression therapy for LBP patients results in increased intervertebral space and reduced disk protrusion (if present) as measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific LBP of at least 6 weeks duration with no evidence of underlying disease or anatomic abnormalities,
* Applicants may have pain radiating to their legs.

Exclusion Criteria:

* Any episode of Acute LBP within the last 6 weeks or less
* Recent Fractures, less than 8 weeks of any bone
* Tumors of any type including soft tissue tumors, myeloma, malignant or documented tumors of any type
* Gross osteoporosis,
* Spondylolisthesis grade 2 and above,
* Hardware fixation, spine fixation or other boney fusion
* Obesity as defined by a BMI greater than 35, body weight over 287 pounds,
* Contra-indication for MRJ assessment,
* Pregnancy,
* neurologic deficits,
* bowel or bladder incontinence,
* progressive lower extremity weakness,
* need for narcotic pain medications for other conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Pain will be measured using a 0-100 visual analog scale. | 19 weeks
Functional activity will be measured using the Roland Morris activity scale | 19 weeks
MRI outcome measures include thickness of disc (disc height, intervertebral space), extent of disc bulging, intervertebral alignment. | 19 weeks

SECONDARY OUTCOMES:
Physical and social activities and quality of life will be measured with the COOP | 19 weeks
Functional health will be measured with the SF-36 | 19 weeks
Depression will be measured using the Geriatric Depression Scale (GDS) | 19 weeks
Treatment satisfaction will be measured using a 5-point Likert scale. | 19 weeks
Reduction in pain medication usage | 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William D Grant, EdD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States